CLINICAL TRIAL: NCT02075398
Title: Evaluation of Respiration Rate Parameters During Motion in Healthy Volunteers Using a Nellcor Bedside Respiratory Patient Monitoring System With Respiration Rate Version 2.0
Brief Title: Nellcor Bedside Respiratory Patient Monitoring System With Respiration Rate Version 2.0
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0428
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2013-12

CONDITIONS: Monitoring Arterial Oxygen Saturation
Keywords: Portable pulse oximeter

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate the Respiration Rate Version 2.0 algorithm, housed in the Nellcor Bedside Respiratory Patient Monitoring System, for performance during motion conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects 18 years or older (inclusive)
* Subject is able to participate for the duration of the study
* Subject is willing to sign an informed consent

Exclusion Criteria:

* Subject with abnormalities that may prevent proper application of the devices
* Physiologic abnormalities that prevent proper application of pulse oximetry sensor
* Severe contact allergies that cause a reaction to standard adhesive materials such as those fund in medical sensors and electrodes
* Subjects with significant arrhythmia, as determined by subject self-report during screening and I/E criteria assessment at study start. (Three events of irregularities in radial pulse with thirty seconds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the available Covidien Boulder Clinical Laboratory subject data base.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the respiration rate performance in healthy adult volunteers during motion when compared to established technologies for measuring parameters related to respiration. | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Scott, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Boulder Clinical Laboratory, Boulder, Colorado, United States